CLINICAL TRIAL: NCT03742908
Title: A Single Center Prospective Randomized Control Trial Investigating the Short-term and Long-term Effects of Intraoperative Prophylactic Antibiotics/Antiseptics on Surgical Outcomes in Chinese Post-mastectomy Breast Reconstruction Patients
Brief Title: Application of Intra-operative Prophylactic Antibiotics/Antiseptics in Chinese Breast Reconstruction Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: E2018124
Record Dates: First submitted 2018-11-07; First posted 2018-11-15 (Actual); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Breast Neoplasms
Keywords: Implant-based breast reconstruction; intraoperative antibiotics/antiseptics; Chinese
MeSH Terms: conditions — Breast Neoplasms | interventions — Cefazolin; Clindamycin

STUDY DESIGN:
Intervention Model Description: Block randomization is generated by one investigator that is not involved in surgery and the block size is kept hidden from other investigators and patients.
Masking Description: Treatment allocation is revealed to the surgical team intraoperatively. Treatment allocation is revealed to the patient post-op in their first followup visit in the clinics.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- saline control (No Intervention): Implant immersion with 100 ml sterile saline (0.9%) for 10 minutes; Breast pocket irrigation (IRRI) with 100ml type III Anerdian for 30 seconds and washed with a total of 1000ml sterile distilled water twice afterwards. No antibiotics is used.
- Cefazolin/clindamycin immersion (Experimental): Implant immersion: implant is immersed with 200mg cefazolin in 100 ml sterile saline (0.9%) for 10 minutes, if the patient is allergic to cefazolin, 600mg clindamycin in 100ml sterile saline (0.9%) is used instead for immersion; Breast pocket irrigation (IRRI) with100ml type III Anerdian for 30 seconds and washed with a total of 1000ml sterile distilled water twice afterwards
  Interventions: Drug: Cefazolin/clindamycin
- Cefazolin/clindamycin immersion+ IRRI (Experimental): Implant immersion: implant is immersed with 200mg cefazolin in 100 ml sterile saline (0.9%) for 10 minutes, if the patient is allergic to cefazolin, 600mg clindamycin in 100ml sterile saline (0.9%) is used instead for immersion; Breast pocket irrigation (IRRI): breast pocket is irrigated with100ml type III Anerdian plus 200mg cefazolin in 100 ml sterile saline (0.9%) for 30 seconds and washed with a total of 1000ml sterile distilled water twice afterwards, if the patient is allergic to cefazolin, 600mg clindamycin in 100ml sterile saline (0.9%) is used instead of cefazolin
  Interventions: Drug: Cefazolin/clindamycin

INTERVENTIONS:
Drug: Cefazolin/clindamycin — Local implant immersion and/or breast pocket irrigation
  Other Names: Ancef; Kefzol; Cleocin
  Arms: Cefazolin/clindamycin immersion; Cefazolin/clindamycin immersion+ IRRI

SUMMARY:
The study aims to investigate different approaches of local application of antibiotics/antiseptics intraoperatively in Chinese patients undergoing post-mastectomy implant based breast reconstruction, and aims to single out an intervention method that limits the use of antibiotics and maintains low rates of surgical site infection and capsular contracture. Patients who undergo post mastectomy breast reconstruction in the breast reconstruction department in Tianjin Medical University Cancer Institute and Hospital are eligible to enter the study.

DETAILED DESCRIPTION:
There is an ongoing trend towards implant based breast reconstruction in post-mastectomy patients in China. In 2015, more than 60% of patients undergoing breast reconstruction in Tianjin Medical University Cancer Institute and Hospital opted for implant based breast reconstruction. One of the major complications in implant based breast reconstruction is infection, which could cause implant explantation, delay the time to adjuvant therapies in breast cancer patients, and inflict adverse psychological effects. Although empirical intravenous and/or oral antibiotics are suggested peri-operatively, local applications of antibiotics/antiseptics and their combinations are applied differently in many medical centers worldwide, and some even suggest against the use of intraoperative local antibiotics. Furthermore, there is no consensus as to the local application of antibiotics intraoperatively for breast reconstruction patients in Chinese population. We therefore designed an open-label prospective randomized control trial in our Chinese patient population to investigate the effects of three different approaches of intraoperative surgical site intervention with antibiotics and or antiseptics. In each groups, all peri-operative interventions are standardized to best reduce bias. Short-term infection rate and long-term capsular contracture rate will be observed in the hope of singling out the best modality in our medical center to integrate into the overall comprehensive treatment for female breast cancer patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent mastectomy and eligible for implant-based breast reconstructions
* Karnofsky Performance Status (KPS) larger than 70
* No severe deficiency in hematological, cardiovascular system, no immunodeficiency, no severe abnormal liver or kidney function

Exclusion Criteria:

* Metastatic breast cancer
* Local or systemic infection within 30 days prior to breast reconstruction surgery
* Local, oral or systemic administration of any form of antibiotics within 30 days prior to breast reconstruction surgery
* Pre-operative complete blood count shows white blood cell (WBC) count >10*10^9/L, Neutrophil cell (N) count > 7.5*10^9/L or N%>80%
* Pre-operative blood procalcitonin (PCT) higher than upper limit of the normal range
* Past history with injection breast augmentation

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female patients with natural breasts
Enrollment: 291 (Estimated)
Dates: Start 2018-06-16 (Actual); Primary Completion 2021-10-31 (Estimated); Study Completion 2021-10-31 (Estimated)

PRIMARY OUTCOMES:
Occurrence of minor surgical site infection | assessed up to 3 months post-op
  the reconstructed breasts present with redness, edema, pain and rise in skin temperature by observation, drainage or wound secretion microbiology culture are positive, the symptoms are relieved by oral antibiotics.
Occurrence of major surgical site infection | assessed up to 3 months post-op
  the reconstructed breasts present with redness, edema, pain and rise in skin temperature by observation, drainage or wound secretion microbiology culture are positive, the symptoms are relieved by intravenous antibiotics or demand surgical interventions such as explantation or change of implant.
Occurrence of capsular contracture | assessed from 3 months post-op up to 2 years post-op or until the trial ends, whichever comes first
  Hardness, pain, and or changes of shape/volume of the reconstructed breasts both by observation or inspected by breast imaging .The grade of capsular contracture is recorded in baker's grading(I-IV).

SECONDARY OUTCOMES:
Occurrence of flap necrosis | assessed up to 1 months post-op
  Complete or partial flap necrosis at the surgical site by surgeon's observation;
Occurrence of hematoma | assessed up to 72 hours post-op
  Peri-prosthetic hematoma observed by hematic drainage and reduced Hematocrit count comparing to normal range;
Occurrence of peri-prosthetic seroma | from 3 months post-op up to 2 years post-op or until the trial ends
  Peri-prosthetic seroma observed by clinical inspection and/or breast imaging;
Baseline and changes of patient's evaluation | evaluate at 6 months as baseline, repeated evaluation at 12 months and 24 months post-op or until the trial ends, whichever comes first, to record changes
  Patient oriented aesthetic and overall satisfaction evaluation using Breast-Q questionnaires (implant reconstructive module)

CONTACTS AND LOCATIONS:
Overall Officials: Jian Yin, Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data (IPD) available to other researchers

REFERENCES:
- [Background] Kummerow KL, Du L, Penson DF, Shyr Y, Hooks MA. Nationwide trends in mastectomy for early-stage breast cancer. JAMA Surg. 2015 Jan;150(1):9-16. doi: 10.1001/jamasurg.2014.2895. PMID 25408966
- [Background] Piper ML, Roussel LO, Koltz PF, Wang F, Singh K, Chin R, Sbitany H, Langstein HN. Characterizing infections in prosthetic breast reconstruction: A validity assessment of national health databases. J Plast Reconstr Aesthet Surg. 2017 Oct;70(10):1345-1353. doi: 10.1016/j.bjps.2017.05.004. Epub 2017 May 18. PMID 28619483
- [Background] Constantine RS, Constantine FC, Rohrich RJ. The ever-changing role of biofilms in plastic surgery. Plast Reconstr Surg. 2014 Jun;133(6):865e-872e. doi: 10.1097/PRS.0000000000000213. PMID 24867746
- [Background] Rubino C, Brongo S, Pagliara D, Cuomo R, Abbinante G, Campitiello N, Santanelli F, Chessa D. Infections in breast implants: a review with a focus on developing countries. J Infect Dev Ctries. 2014 Sep 12;8(9):1089-95. doi: 10.3855/jidc.3898. PMID 25212072
- [Background] Reish RG, Damjanovic B, Austen WG Jr, Winograd J, Liao EC, Cetrulo CL, Balkin DM, Colwell AS. Infection following implant-based reconstruction in 1952 consecutive breast reconstructions: salvage rates and predictors of success. Plast Reconstr Surg. 2013 Jun;131(6):1223-1230. doi: 10.1097/PRS.0b013e31828bd377. PMID 23714788
- [Background] Alderman A, Gutowski K, Ahuja A, Gray D; Postmastectomy ExpanderImplant Breast Reconstruction Guideline Work Group. ASPS clinical practice guideline summary on breast reconstruction with expanders and implants. Plast Reconstr Surg. 2014 Oct;134(4):648e-655e. doi: 10.1097/PRS.0000000000000541. PMID 25357060
- [Background] Barr SP, Topps AR, Barnes NL, Henderson J, Hignett S, Teasdale RL, McKenna A, Harvey JR, Kirwan CC; Northwest Breast Surgical Research Collaborative. Infection prevention in breast implant surgery - A review of the surgical evidence, guidelines and a checklist. Eur J Surg Oncol. 2016 May;42(5):591-603. doi: 10.1016/j.ejso.2016.02.240. Epub 2016 Feb 27. PMID 27005885
- [Background] Phillips BT, Fourman MS, Bishawi M, Zegers M, O'Hea BJ, Ganz JC, Huston TL, Dagum AB, Khan SU, Bui DT. Are Prophylactic Postoperative Antibiotics Necessary for Immediate Breast Reconstruction? Results of a Prospective Randomized Clinical Trial. J Am Coll Surg. 2016 Jun;222(6):1116-24. doi: 10.1016/j.jamcollsurg.2016.02.018. Epub 2016 Mar 4. PMID 27106640
- [Background] Phillips BT, Halvorson EG. Antibiotic Prophylaxis following Implant-Based Breast Reconstruction: What Is the Evidence? Plast Reconstr Surg. 2016 Oct;138(4):751-757. doi: 10.1097/PRS.0000000000002530. PMID 27307337
- [Background] Huang N, Liu M, Yu P, Wu J. Antibiotic prophylaxis in prosthesis-based mammoplasty: a systematic review. Int J Surg. 2015 Mar;15:31-7. doi: 10.1016/j.ijsu.2015.01.020. Epub 2015 Jan 29. PMID 25638736
- [Background] Gowda AU, Chopra K, Brown EN, Slezak S, Rasko Y. Preventing Breast Implant Contamination in Breast Reconstruction: A National Survey of Current Practice. Ann Plast Surg. 2017 Feb;78(2):153-156. doi: 10.1097/SAP.0000000000000822. PMID 27464530
- [Background] Frois AO, Harbour PO, Azimi F, Young J, Chan B, Mak C, Warrier S. The Role of Antibiotics in Breast Pocket Irrigation and Implant Immersion: A Systematic Review. Plast Reconstr Surg Glob Open. 2018 Sep 14;6(9):e1868. doi: 10.1097/GOX.0000000000001868. eCollection 2018 Sep. PMID 30349776